CLINICAL TRIAL: NCT03004235
Title: ED Data Collection of Suspected Carbon Monoxide Poisoning
Brief Title: Suspected Cases of Carbon Monoxide Poisoning in the ED
Status: Terminated | Type: Observational
Why Stopped: IRB is reviewing all studies at the institution and are on hold
Sponsor: Nonin Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: QATP2978
Record Dates: First submitted 2016-12-21; First posted 2016-12-28 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2018-07

CONDITIONS: Carbon Monoxide Poisoning
MeSH Terms: conditions — Carbon Monoxide Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Observational data collection — Observational data collection

SUMMARY:
The purpose of this study is to collect non-invasive observational data in suspected or known carbon monoxide poisoning.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected carbon monoxide poisoning

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be selected based on symptoms in the Emergency Department.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2016-12; Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Values from the test device will be compared to the values from co-oximetry to determine the accuracy of the test device | Through study completion, an average of 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: James Miner, MD, Principal Investigator — Hennepin County Medical Center, Minneapolis
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No